CLINICAL TRIAL: NCT05893511
Title: Upfront Endoscopic Ultrasound-guided Gallbladder Drainage (EUS-GBD) Versus Standard Protocol (Antibiotics First) for Mild to Moderate Acute Cholecystitis in Patients Who Are Very-high-risk for Cholecystectomy: A Randomized-controlled Trial.
Brief Title: EUS-GBD vs Antibiotics for Patients at High Risk for Cholecystectomy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CHAN SHANNON MELISSA, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022.518
Record Dates: First submitted 2023-03-27; First posted 2023-06-08 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Acute Cholecystitis
Keywords: acute cholecystitis; EUS-guided gallbladder drainage; antibiotics
MeSH Terms: conditions — Cholecystitis, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antibiotics first group (Active Comparator): Antibiotics first equals to intravenous antibiotics 2nd generation cephalosporin or equivalent). Antibiotics would first be given parenterally and then switched to oral form when patient can tolerate diet or when sepsis subside. It will be continued for at least a total of 7 days.
  Interventions: Drug: Antibiotics first
- Endoscopic ultrasound-guided gallbladder drainage (EUS-GBD) (Active Comparator): Prior to the procedure, the patients would be kept fasted for 6 hours and antibiotics would be commenced (2nd generation cephalosporin or equivalent). Antibiotics would be continued for up to one week after the procedure.EUS-GBD would be performed by either the conventional or direct method.
  Interventions: Procedure: Endoscopic ultrasound-guided gallbladder drainage

INTERVENTIONS:
Procedure: Endoscopic ultrasound-guided gallbladder drainage — Prior to the procedure, the patients would be kept fasted for 6 hours and antibiotics would be commenced (2nd generation cephalosporin or equivalent). EUS-GBD would be performed by either the conventional or direct method. A 10mm stent system would be used if the largest gallstone is smaller than 10mm in size and a 16mm stent is used if the largest gallstone is larger than 10mm. The distal flange of the stent would be deployed under EUS guidance, followed by deployment of the proximal flange under endoscopic guidance. Once deployed, the gallbladder is completely emptied by suction and irrigation until the effluent through the stent is clean. The need of inserting an additional double pigtail plastic stent through the LAMS would be decided by the endosonographer. A course of antibiotics will be continued for 7 days after the procedure .
  Arms: Endoscopic ultrasound-guided gallbladder drainage (EUS-GBD)
Drug: Antibiotics first — Patients randomized to antibiotics first would be given intravenous antibiotics 2nd generation cephalosporin or equivalent). Antibiotics would first be given parenterally and then switched to oral form when patient can tolerate diet or when sepsis subside. It will be continued for at least a total of 7 days.
  Arms: Antibiotics first group

SUMMARY:
Objectives Acute cholecystitis commonly occurs in elderly patients who are at high-risk for surgery. Whether upfront Endoscopic ultrasound-guided gallbladder drainage (EUS-GBD) is advantageous over antibiotics first for mild acute cholecystitis is uncertain.

Hypothesis to be tested The aim is to compare EUS-GBD versus standard protocol (antibiotics first) as a definitive treatment, in very high-risk patients suffering from mild to moderate acute cholecystitis. We hypothesize that EUS-GBD can reduce the 1-year risk of recurrent acute cholecystitis.

Design and subjects This is an international randomised controlled study including consecutive patients suffering from acute cholecystitis that are very high-risk for cholecystectomy. The patients would be randomized to receive EUS-GBD or antibiotics first.

Interventions: EUS-GBD versus antibiotics

Main outcome measures:

The primary outcome is the rate of recurrent acute cholecystitis in 1 year. Other outcomes include technical and clinical success, post-procedural pain scores, analgesic requirements, adverse events, re-admissions, re-interventions, quality of life and cost analysis.

Data analysis All outcomes would be analysed according to the intention-to-treat principle. Kaplan-Meier method with the log-rank test will be used to compare differences in recurrent acute cholecystitis in 1 year. A health economic analysis will also be performed. Assuming a 17.1% difference in recurrent acute cholecystitis rates, a 2-sided P value of 0.05, a power of 80%, and a 10% dropout rate, 110 patients is required.

Expected results The findings of this study can help establish the role of EUS-GBD in management of high-risk patients suffering from acute cholecystitis over antibiotics alone and Percutaneous transhepatic gallbladder drainage.

ELIGIBILITY:
Inclusion Criteria:

1. Consecutive patients aged ≥ 18 years old
2. Suffering from grade 1 or 2 acute calculous cholecystitis*
3. At very high-risk for early laparoscopic cholecystectomy due to poor premorbid conditions** or elderly patients suffering from acute cholecystitis but refused operations

Exclusion Criteria:

Patients with the following conditions are excluded from the study:

* Pregnancy
* Patients unwilling to undergo follow-up assessments
* Patients with suspected gangrene or perforation of the gallbladder
* Grade III acute cholecystitis33
* Patients diagnosed with concomitant liver abscess or pancreatitis (defined as elevated serum amylase more than three times the upper limit of normal)
* Altered anatomy of the upper gastrointestinal tract due to surgery of the esophagus, stomach and duodenum
* Patients with liver cirrhosis, portal hypertension and/or gastric varices
* Abnormal coagulation: International normalized ratio (INR) > 1.5 and/or platelets < 50.000/mm3
* Previous drainage of the gallbladder
* Patients suffering acute cholecystitis due to malignant cystic duct obstruction
* Patients with life expectancy of less than 3 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-04-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
1-year recurrent acute cholecystitis rate | 1-year
  recurrent acute cholecystitis rate in 1 year

SECONDARY OUTCOMES:
Technical success | 1-year
  Technical success is defined as the ability to access and drain the gallbladder by placement of a drainage tube or maintenance of good drainage.
Daily post-procedural pain scores for the first 7 days | 7 days
  Pain assessment would be performed using the visual-analogue scale (1 to 100) on post-procedural days 1 to 7.
Type and dosage of analgesic required | an average of 7 days
  Type and the dosage of the analgesic required after procedure/administered of antibiotics would be recorded.
Adverse events | 1-year
  Any adverse events occured in 1 year will be recorded
Total number of unplanned readmissions related to acute cholecystitis and reinterventions | 1-year
  The total number and the reason of any unplanned readmissions related to acute cholecystitis and reinterventions in 1 year will be recorded.
Cost-effectiveness measurement | 1-year
  1. All costs in the antibiotics first arm would be recorded: the cost of using antibiotics (dose, frequency, duration), the cost of Percutaneous Transhepatic Gallbladder Drainage (PT-GBD) and subsequent cholecystogram if any
  2. All costs in the EUS-GBD arm would be recorded: the cost of EUS-GBD procedure (including the procedure itself, anaesthesia, Lumen-apposing metal stents (LAMS), needle, guidewire), cost of managing complications if any
  3. All costs in both arms would be recorded:
  i. Index admission: the cost of investigations (blood test, imaging), medications, hospital stay ii. Unplanned readmissions: the cost of investigations, medications, reinterventions (cost of procedure and its equipment) iii. Cost of the follow-up clinic visits
Quality of life assessment | 1-year
  EQ-5D on admission (before randomisation) and at every follow-up clinic visit
Clinical success (clinical symptoms) | 1-year
  Clinical success is defined as afebrile on post-treatment day 3, or temperature downward trend; and resolution of peritoneal signs.
Clinical success (laboratory tests) | 1-year
  Clinical success is defined as leucocytes count of >=30% drop on post-treatment Day 3 or normalised.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Melissa Chan, Principal Investigator — The Chinese Universtiy of Hong Kong
Locations (1):
- The Chinese Universtiy of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No